CLINICAL TRIAL: NCT04738734
Title: A Multicenter, Prospective, Randomized, Comparison IDE Study Between the Pulse Biosciences CellFX System and Cryosurgery for the Treatment of Cutaneous Non-Genital Common Warts
Brief Title: CellFX Comparison to Cryosurgery in Cutaneous Non-Genital Common Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP-WC-015
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Warts; Warts Hand; Verruca
Keywords: CellFX; Nano-Pulse Stimulation; NPS; Clearance; Wart Reduction
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Each subject will be evaluated by the blinded site investigator conducting assessment of outcomes at 7, 30, 60, and 90-days following CellFX and Cryosurgical treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- CellFX Procedure (Experimental): CellFX device using pre-defined energy protocols
  Interventions: Device: CellFX System Device
- Cryosurgical Procedure (Active Comparator): Cryosurgery will be standardized across all investigational sites. Investigators will perform the Cryosurgical procedure using the Brymill Cry-Ac B700 Liquid Nitrogen Sprayer.
  Interventions: Device: Cryosurgery Liquid Nitrogen Sprayer

INTERVENTIONS:
Device: CellFX System Device — The CellFX System utilizes non-thermal, localized delivery of a timed series of low energy, nanosecond electrical pulses that can trigger regulated cell death.
  Arms: CellFX Procedure
Device: Cryosurgery Liquid Nitrogen Sprayer — Cryosurgery will be standardized across all investigational sites using the Brymill Cry-Ac spray canister with standard cryoprobe.
  Arms: Cryosurgical Procedure

SUMMARY:
This prospective, multicenter, single-blinded, randomized comparison study is designed to compare the safety and effectiveness of the CellFX System to Cryosurgery for the clearance of cutaneous non-genital common warts on all areas of the body excluding the scalp, nose, within the orbital region of the face, plantar or periungual area in healthy adult subjects.

DETAILED DESCRIPTION:
The study will enroll healthy adult subjects with a minimum of two cutaneous non-genital warts, excluding the face, with each wart lesion not exceeding 10 x 10mm. Macrophotography of all study warts will be captured along with a blinded site Investigator to characterize wart healing, wart clearance and wart reduction. All subjects will be followed at 7, 30, 60, and 90-days following the last CellFX or Cryosurgical Procedure. All wart lesions are eligible for up to a total of 3 treatments over the course of the study. Adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 21 and not older than 80 years of age
* Subject has a Fitzpatrick Skin Type I, II, III or IV.
* Subject gives voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subject must comply with study procedures including all follow-up visits.
* Subject is willing to have warts treated in a single treatment session and understands that their warts may undergo multiple treatment sessions at subsequent visits.
* Subject must have a minimum of 2 warts and up to 8 warts to be treated.
* Subject with a clinical diagnosis of common warts located on hands and fingers or other body areas that are not located on the scalp, nose, within the orbital region of the face, plantar, genital or periungual area.
* For study purposes, the warts must be no greater than 3 mm in height and must not exceed 10mm x 10mm at their largest dimension.
* Each wart must appear alone and discrete and not appear in clusters.
* Each wart must have been present for at least 4 weeks.
* Subject consents to have photographs taken of the warts.
* Subject agrees to refrain from using all other wart removal products or treatments (e.g.

topical medication including over-the-counter medications) during the study period.

Exclusion Criteria:

* Subject with more than 8 visible warts in total anywhere on the body.
* Subject has flat, periungual, subungual, genital, anal, mosaic, plantar or filiform warts.
* Subject has an implantable electronic medical device.(i.e., pacemaker, implantable cardioverter defibrillator)
* Subject has an active infection or history of infection in designated test area within 90 days prior to first treatment.
* Subject is taking antihistamines, including those used for gastric symptoms.
* Subject is prone to Koebnerization or has any of the following conditions (e.g., psoriasis, vitiligo, lichen planus, or an autoimmune disorder of the skin)
* Subject is not willing or able to sign the Informed Consent.
* Subject is known to be immune compromised.
* Subject has allergies to Lidocaine or Lidocaine-like products.
* Subject is a member of a vulnerable population including individuals employed by the
* Sponsor, clinic site, or entity associated with the conduct of the study.
* Have any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study.
* Use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study.
* Subject was previously treated with CellFX for warts.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (10):
- United States (10):
  - Investigate MD, Scottsdale, Arizona
  - Moy-Fincher-Chipps Dermatology, Beverly Hills, California
  - AboutSkin Dermatology and DermSurgery, Greenwood Village, Colorado
  - Palm Harbor Dermatology, Clearwater, Florida
  - Oak Dermatology, Joliet, Illinois
  - Juva Skin & Laser Center, New York, New York
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Austin Institute for Clinical Research, Inc., Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CellFX Procedure | Cryosurgical Procedure
Started | 75 | 75
Completed | 68 | 67
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 5 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Mistake of termination of subject by clinical site | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CellFX Procedure | Cryosurgical Procedure | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Full Range); unit: Years] | 44.6 [18 to 78] | 46.2 [18 to 80] | 45.4 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 44 | 80
  Male | 39 | 31 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 68 | 65 | 133
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 70 | 67 | 137
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 3 | 3
Warts [Number; unit: warts] — Total number of enrolled warts per treatment
  warts | 231 | 248 | 479

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Warts Resolved
Description: The primary effectiveness endpoint is the percentage of warts resolved or cleared as assessed "live" by the blinded site investigator at 30 days after the last treatment with CellFX or Cryosurgical Procedure.
Time Frame: 30 days following the last CellFX or Cryosurgical Procedure up to a maximum of 3 months
Population: The population consisted of participants with treated warts and evaluated at 30-days following the last CellFX or Cryosurgical Procedure up to a maximum of 3 months.
Measure: Mean (95% Confidence Interval); unit: percentage of warts resolved
Units Other Than Participants: wart lesions
Arm/Group | CellFX Procedure | Cryosurgical Procedure
Number analyzed (Participants) | 70 | 69
Number analyzed (wart lesions) | 216 | 232
percentage of warts resolved | 80.7 [71.1 to 90.2] | 73.1 [64.2 to 81.9]

2. Primary Outcome: Percentage of Warts Treated With Skin Textural Changes
Description: The safety endpoint is the percentage of warts with skin textural changes where the wart was originally treated and showed textual changes of the surrounding skin where the wart was treated and included; scabbing, swelling, crusting, blister, or ulceration when assessed by the blinded site investigator.
Time Frame: 30 days from the last CellFX or Cryosurgical Procedure up to a maximum of 3 months
Population: The population consisted of participants with treated warts and evaluated for skin textural changes at 30-days following the last CellFX or Cryosurgical Procedure up to a maximum of 3 months.
Measure: Mean (95% Confidence Interval); unit: percentage of warts
Units Other Than Participants: wart lesions
Arm/Group | CellFX Procedure | Cryosurgical Procedure
Number analyzed (Participants) | 70 | 69
Number analyzed (wart lesions) | 216 | 232
percentage of warts | 41.4 [32.5 to 50.3] | 13.1 [5.73 to 20.5]

3. Primary Outcome: Presence of Pigmentary and Scarring Skin Changes
Description: The skin change safety event is defined as the presence of hyperpigmentation, hypopigmentation, or scarring as assessed by the blinded site investigator.
Time Frame: 90 days from the last CellFX or Cryosurgical Procedure up to a maximum of 6 months
Population: The population consisted of participants with treated warts and evaluated at 90-days following the last CellFX or Cryosurgical Procedure up to a maximum of 6 months.
Measure: Mean (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: wart lesions
Arm/Group | CellFX Procedure | Cryosurgical Procedure
Number analyzed (Participants) | 68 | 67
Number analyzed (wart lesions) | 208 | 227
percentage of lesions | 37.3 [25.5 to 49.0] | 23.7 [14.1 to 33.3]

ADVERSE EVENTS:
Time Frame: 150 days
Arm/Group | CellFX Procedure | Cryosurgical Procedure
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 10/75 | 2/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CellFX Procedure (N=75) | Cryosurgical Procedure (N=75)
Skin Neoplasm (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) — Presence of non-melanoma skin cancer (SCC) was at the site of the treated lesion along with an Actinic Keratotic lesion treated with Cryotherapy. One participant showed a BCC lesion not related to treatment site.
Neoplasm of uncertain behavior of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Biopsy showed wart
Paraesthesia (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) — Numbness or altered sensation at the site of treatment
Neuropathy (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Sensory disturbance including numbness or altered sensation and resolved within 2-6 days
Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Suspect Skin Infection, no culture collected
Tinea Versicolor (Infections and infestations) | 1 (1) | 0 (0) — Participant has recurrent fungal infections that usually have resolved within 2 months.
Pain (General disorders) | 2 (2) | 0 (0) — Post-procedure pain for one participant that resolved less than 24 hours. Second participant had persistent pain post treatment that resolved within 5 months without intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT04738734/Prot_SAP_000.pdf